

## NON-INTERVENTIONAL STUDY PROTOCOL STUDY INFORMATION

| Title | Patient characteristics, treatment patterns and incidence of events (discontinuation, persistence, key primary clinical outcomes) in NVAF patients initiating OAC therapy in Colombia |
|---|---|
| Protocol number | B0661148 |
| Protocol version identifier | 1.0 |
| Date of last version of protocol | 10 October 2019 |
| Active substance | Apixaban |
| Medicinal product | Eliquis |
| Research question and objectives | <ul> <li>To assess demographic and clinical characteristics of NVAF patients treated with Oral Anticoagulants (OACs) in Colombia.</li> <li>To describe treatment patterns (eg OAC usage, dose, concomitant medications, persistence)</li> <li>Exploratory Objectives</li> <li>To descriptively assess the time to clinical events (Effectiveness and Safety Outcomes) among patients persistent on OAC therapy</li> <li>Effectiveness outcomes: First stroke/ Systemic Embolism;</li> <li>Safety outcomes: Major bleeding,</li> </ul> |
| Author | PPD PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

#### TABLE OF CONTENTS

| LIST OF ABBREVIATIONS | |
|---|---|
| 1. RESPONSIBLE PARTIES | ······································ |
| 2. ABSTRACT | |
| 3. AMENDMENTS AND UPDATES | |
| 4. MILESTONES | |
| 5. RATIONALE AND BACKGROUND | |
| 6. RESEARCH QUESTION AND OBJECTIVES | 14 |
| 7. RESEARCH METHODS | 15 |
| 7.1. Study Design | 15 |
| 7.2. Setting | |
| Inclusion Criteria | |
| Exclusion Criteria | |
| 7.2.3. Cohorts | |
| 7.3. Variables | |
| Definition of outcome variables | 23 |
| 7.4. Data Sources | 44 |
| 7.4.1. Claim Database | 44 |
| 7.4.2. Medical Record | 44 |
| 7.5. Study Size | 44 |
| 7.6. Data Management | 44 |
| 7.6.1 Electronic Case Report (ECR) | 44 |
| 7.6.2 Record Retention | 45 |
| 7.6.3 Patient Identification | 40 |
| 7.6.4 Collection of Information | 40 |
| 7.6.5 Database Retention | 40 |
| 7.7 Data Analysis | 40 |
| 7.7.1 Missing Data Management | 4 |
| 7.8 Quality Control | |
| 7.9 Limitations of the research methods | 4 |
| 7.10 Other aspects | 48 |
| 8 PROTECTION OF STUDY SUBJECTS | |
| 8.1 Patient Information | |
| 8.2 Patient Consent | 48 |
| 8.4 Ethical Conduct of the Study | |
| ř | |
| 9 MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 50 |
| 10 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 51 |
| 11. REFERENCES | 52 |
| 12. LIST OF TABLES | 53 |
| 13. LIST OF FIGURES | 53 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 53 |
| ANNEX 2 ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 53 |

| Apixaban |
|---------------------------------------------|
| B0661148- NON-INTERVENTIONAL STUDY PROTOCOL |
| Final, 10 October 2019 |
| ANNEY 3 ADDITIONAL INFORMATION |

#### LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ARB | Angiotensin II receptor blockers |
| ACE | Angiotensin-converting-enzyme inhibitor |
| AE | Adverse event |
| AEM | Adverse event monitoring |
| AIDS | Acquired Immune Deficiency Syndrome |
| AF | Atrial fibrillation |
| ANOVA | Analysis of variance |
| ATC | Anatomical Therapeutic Chemical |
| | C: Congestive heart failure |
| | H: Hypertension |
| | A: Age ≥75 years |
| | D: Diabetes mellitus |
| CHA <sub>2</sub> DS <sub>2</sub> -VASc | S <sub>2</sub> : Prior Stroke or transient ischemic attack or Thromboembolism |
| | V: Vascular disease (peripheral artery disease, myocardial infarction, aortic |
| | plaque) |
| | A: Age 65–74 years |
| | Sc: Sex category ( female sex) |
| | C: Congestive heart failure |
| | H: Hypertension |
| $CHADS_2$ | A: Age ≥75 years |
| _ | D: Diabetes mellitus |
| | S <sub>2</sub> : Prior Stroke or transient ischemic attack or Thromboembolism |
| COPD | Chronic obstructive pulmonary disease |
| ECR | Electronic Case Report |
| GEP | Good Epidemiological Practice |
| GPP | Good Pharmacoepidemiology Practices |
| GII | H: Hypertension |
| | A: Abnormal renal and liver function |
| | S: Stroke |
| HAS-BLED | B: Bleeding |
| In to BEEB | L: Labile INR |
| | E: Elderly |
| | D: Drugs or alcohol |
| НМО | Health Maintenance Organizations |
| ICD-10 | 10th revision of the International classification of diseases |
| IEA | International Epidemiological Association |
| IEC | Independent Ethics Committee |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| ISPE | International Society for Pharmacoepidemiology |
| ISPOR | International Society for Pharmacoeconomics and Outcomes Research |
| MANOVA | Multivariate analysis of variance |
| NI | Non- interventional |
| NIS | Non-interventional study |
| NOAC | New oral anticoagulant |
| NSAID | Non-steroidal anti-inflammatory drugs |
| NVAF | Non-valvular atrial fibrillation |
| 117711 | 11011 Tell deller Holliedon |

# Apixaban B0661148- NON-INTERVENTIONAL STUDY PROTOCOL Final, 10 October 2019

| Abbreviation | Definition |
|---|---|
| OAC | Oral anticoagulant |
| | S: Sex (female) |
| | A: Age (<60 years) |
| CAMA TT D | Me: Medical history |
| SAMe-TT <sub>2</sub> R <sub>2</sub> | T: Treatment |
| | T: Tobacco use (within 2 years) |
| R: Race (non-Caucasian) | |
| SPSS | Statistical Package for the Social Sciences |
| TIA | Transient ischaemic attack |
| VKA | Vitamin K Antagonist |
| VTE | Venous thromboembolism |

#### 1. RESPONSIBLE PARTIES

This document contains information that is confidential and proprietary to the sponsor. This information is being provided to you for the purposes of study evaluation or conduction. The contents of this study may only be disclosed to your review board, ethics committees or regulatory agencies under confidential conditions. The contents of this document may not be used in any other study, disclosed to other persons or entities, or published without authorization from the sponsor. Any other information which might be added to this document is also confidential and proprietary to the sponsor following the same considerations of this document.

#### **Principal Investigator of the Protocol**

| Name, degree(s) | Job Title | Affiliation | Address |
|-----------------|-----------|-------------|---------|
| PPD | MD, MSc | PPD | PPD |
| MD | | | |

**Country Coordinating Investigators** 

| Country Coordinating Investigators | | | |
|---|---|---|---|
| Name, degree(s) | Job Title | Affiliation | Address |
| PPD | MD, MSc | PPD | PPD |
| PPD MD, MSc | · | | PPD |
| PPD | MD, MSc | PPD | PPD<br>PPD |
| PPD | Pharmacist, MSc | PPD | PPD<br>PPD |
| PPD | Economist | PPD | PPD |
| | | | PPD |

#### 2. ABSTRACT

| <b>Study title:</b> Patient characteristics, treatment patterns and incidence of events (discontinuation, persistence, | | | | | | |
|---|---|---|---|---|---|---|
| key primary clinical outcomes) in NVAF patients initiating OAC therapy in Colombia | | | | | | |
| Protocol number | B0661148 | Phase | 4 | Type | | Observational |
| Condition/Disease | Non-valvular atrial | fibrillation | (N | (VAF) | | |
| Number of patients | The total population | | | <b>Duration of</b> | | ow-up will be performed |
| | patients treated with | ı OAC | | the patients | until | the patient presents a |
| | between January 1, | 2013 and | | in the study | swite | ch, discontinuation, death, |
| | June 30, 2018 was analyzed in | | | | even | t of stroke / systemic |
| | the claim dabtabase. For the | | | | emb | olism or major bleeding, |
| | purpose of the study, it | | | | or ur | ntil June 30, 2019. |
| | contains the inform | | | | | |
| | 7,500 patients, once they were | | | | | |
| | verified that they met the | | | | | |
| | inclusion criteria of the study. | | | | | |
| | | • | | | | |
| Country participants | Colombia | | | <b>Duration of</b> | 8 mc | onths |
| | | | | the study | | |

#### Rational and background:

Non-valvular atrial fibrillation (NVAF) is an acute or chronic heart disorder that is associated with an increase in the mortality rate, strokes and other thromboembolic events (1). This is further increased by individual conditions of patients, such as hypertension, abnormal renal or hepatic function, stroke, history of or predisposition to bleeding, people over 65, among others. (2)

One of the standard treatments for management of these patients is usually vitamin K antagonists (VKA, for example, warfarin); in the analysis of net clinical benefits of this therapy it is suggested that the effect of VKA is even more positive in patients with a high score on the HAS-BLED (hypertension, abnormal renal/liver function, stroke, bleeding history or predisposition, labile International Normalized Ratio, elderly, drugs/alcohol concomitantly) scale. (3) Another therapeutic alternative is the new oral anticoagulants (NOACs) — dabigatran, rivaroxaban and apixaban —, which according to evidence have advantages in efficacy and safety compared to warfarin (4) and even when the risk of bleeding and stroke are high, the net clinical benefit appears to be greater when compared to warfarin. (5) Likewise, there is a lower prevalence of intracranial hemorrhage and its different subtypes of patients being treated with new oral anticoagulants when compared to warfarin. (6)

While it is true there are several studies that seek to understand the characteristics of patients who were diagnosed with NVAF under different treatment options, and even subpopulation analyses, the evidence at the national level is limited, both in demographic and clinical characteristics and in treatment patterns of this population. In a retrospective descriptive study of an emergency department in a third level care center in the city of Bogota, it was observed that the main comorbidities of patients with atrial fibrillation (AF) were arterial hypertension and heart failure where most patients do not receive anticoagulation. (7) In turn, for the overall population it is estimated that the prevalence of AF in Colombia (4.8%) seems to be higher than that reported in developed countries (0.03% to 1.25%) (8), according to a study conducted in a university hospital in the country (9).

Taking into account the limited knowledge on the use of oral anticoagulants in patients diagnosed with NVAF in the country and, even more in the differences in the response to these therapies in different patient subpopulations. The purpose of this study is to assess the demographic and clinical characteristics, treatment patterns and incidence of events (discontinuation, persistence, key primary clinical outcomes) in NVAF patients that initiated OACs in study period.

#### Primary Objectives

- To assess demographic and clinical characteristics of NVAF patients treated with oral anticoagulants (OACs) in Colombia.
- To describe treatment patterns (eg OAC usage, dose, concomitant medications, persistence)

#### **Exploratory Objectives**

• To descriptively assess the time to clinical events (Effectiveness and Safety Outcomes) among patients persistent on OAC therapy

Effectiveness outcomes: First Stroke/ Systemic Embolism; CCI
Safety outcomes: Major bleeding CCI

#### Design:

Observational, descriptive study of a retrospective cohort of adult patients diagnosed with NVAF in selected Health Maintenance Organizations (HMO) of Colombia. These patients will be identified from the drug claim database, whose index date of the study will be the first prescription with any of the oral anticoagulants, that is, they are patients with NVAF for the first time starting a therapy with any of the NOACs between January 1, 2013 and June 30, 2018 and follow up period will be among January 2013 to July 2019, to ensure that the last patients can provide follow-up for one year. Patients will be required to have an NVAF diagnosis before or on the index date and health plan for 6 months pre-index date (baseline period).

#### Population:

The total population of patients treated with any oral anticoagulant between January 1, 2013 and June 30, 2018 will be analyzed in the claim database. This means that patients who start warfarin and NOACs would be included within this period. Patients who initiate NOACs within the established period and who have been exposed to warfarin before 2013 will also be included.

#### **Inclusion criteria:**

Patients must meet the following inclusion criteria in order to be able to take part in the study:

- a) Patients with a diagnosis of AF considered according to the following diagnoses as per the 10th revision of the International classification of diseases (ICD-10) I48 codes at some point before or on the index date, without recorded valvular disease;
- b) Patients who have started treatment with apixaban, dabigatran, rivaroxaban and warfarin for the first time during the identification period, understanding as start of drug delivery by insurer, and after the diagnosis of AF between January 1, 2013 to June 30, 2018;
- c) Patients starting apixaban, dabigatran, rivaroxaban from January 1, 2013 to June 30, 2018 in patients previously exposed to warfarin;
- d) Patient had continuous health plan enrolment for 6 months pre-index date (baseline period);
- e) Patients older than 18 years old on the index date;
- f) NVAF diagnosis before or on the index date.

#### **Exclusion criteria:**

Patients who meet any of the following criteria will not be included in the study:

- a) Patients with any of the following diagnoses prior to the use of the treatments of interest or index date:
  - Valvular heart disease or valve replacement ICD-10 codes: I05, I06, I07, I08, I09, I21, I22, I34, I35, I36, I37, I38, I39, I700, I702-I709; Q22, Q23, Q25, T82, Z95
  - Pregnancy during the study period. ICD-10 O00-O9A
  - Diagnosis of venous thromboembolism (VTE) ICD-10 codes: I26, I80 I82;
- b) Individuals with a transitory diagnosis of NVAF prior to the use of the treatments of interest or index date:
- c) Exposure to more than one OAC on or after the index date, during the follow-up period;
- d) NOAC doses different from those recommended by the manufacturing laboratories.

#### **Data Collection:**

#### Apixaban

#### B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

Final, 10 October 2019

The information will be analyzed in two moments: (i) the period of the index date, where the baseline information of patients will be collected; (ii) and the follow-up period, during this period the clinical results will be evaluated as well as the continuation of the treatment in the study population and for specific subpopulations.

#### Variables:

- Clinical and demographic characteristics
- Treatment patterns (OAC usage, dose, concomitant medications, persistence)

#### **Effectiveness outcomes:**

• First CCI switch of treatment, first event of stroke/ systemic embolism

#### Safety outcomes:

• Major bleeding





#### Data sources:

The information will be used in the study comes exclusively form secondary sources.

- Claim database:
  - The persistence on therapy and treatment patterns (duration of treatment, changes, persistence), pharmacy claim information, demographic information, diagnosis and insurance data.
- Medical records
  - Baseline demographic and clinical characteristics and the information related to the outcomes of interest (stroke/systematic embolism, bleeding events and death)

#### Statistic analysis

This type of analysis is descriptive and explanatory, as it depends largely on the sample size. Continuous variables will be presented as means, standard deviation or other measures of central tendency or position, while categorical variables will be presented as frequencies and percentages.

Regarding bivariate analyses of continuous variables with normal behavior, the Student's t test will be performed. In case of presenting non-normal behavior, the Mann-Withney test will be used. For variables that are continuous with several categories, analysis of variance (ANOVA) will be assessed. In the event of presenting a non-normal behavior, the multivariate analysis of variance (MANOVA) test will be carried out. For categorical variables, the  $X^2$  test will be used.

The cumulative incidence of clinical outcomes (stroke/ systemic embolism and major bleeding) will be calculated throughout the study period, from which the incidence or survival curves will be derived using the Kaplan Meier method. Incidence of events will be explored in clinically relevan subgroups based on sample size.

A similar analysis will be performed for the group of patients who have not presented stroke/ systemic embolism or major bleeding events to estimate the time for discontinuation events and change of treatment.

In the independent variables, the significance will be analyzed, as a level of statistical significance p < 0.05.

### 3. AMENDMENTS AND UPDATES

None

#### 4. MILESTONES

| Milestone | Planned Data |
|--------------------------|-------------------|
| Start of data collection | November 15, 2019 |
| End of data collection | March 31, 2020 |
| Data analysis | CCI |
| Preliminary report | CCI |
| Final study report | CCI |

#### 5. RATIONALE AND BACKGROUND

Non-valvular atrial fibrillation (NVAF) is an acute or chronic heart disorder that is associated with an increase in the mortality rate, strokes and other thromboembolic events (1). This is further increased by individual conditions of patients, such as hypertension, abnormal renal or hepatic function, stroke, history of or predisposition to bleeding, people over 65, among others. (2)

One of the standard treatments for management of these patients is usually vitamin K antagonists (VKA, for example, warfarin); in the analysis of net clinical benefits of this therapy it is suggested that the effect of VKA is even more positive in patients with a high score on the HAS-BLED (hypertension, abnormal renal/liver function, stroke, bleeding history or predisposition, labile International Normalized Ratio, elderly, drugs/alcohol concomitantly) scale. (3) Another therapeutic alternative is the new oral anticoagulants (NOAC) — dabigatran, rivaroxaban and apixaban —, which according to evidence have advantages in efficacy and safety compared to warfarin (4) and even when the risk of bleeding and stroke are high, the net clinical benefit appears to be greater when compared to warfarin. (5) Likewise, there is a lower prevalence of intracranial hemorrhage and its different subtypes of patients being treated with new oral anticoagulants when compared to warfarin. (6)

While it is true there are several studies that seek to understand the characteristics of patients who were diagnosed with NVAF under different treatment options, and even subpopulation analyses, the evidence at the national level is limited, both in demographic and clinical characteristics and in treatment patterns of this population. In a retrospective descriptive study of an emergency department in a third level care center in the city of Bogota, it was observed that the main comorbidities of patients with atrial fibrillation (AF) were arterial hypertension and heart failure where most patients do not receive anticoagulation. (7) In turn, for the overall population it is estimated that the prevalence of AF in Colombia (4.8%) seems to be higher than that reported in developed countries (0.03% to 1.25%) (8), according to a study conducted in a university hospital in the country (9).

Taking into account the limited knowledge on the use of oral anticoagulants in patients diagnosed with NVAF in the country and, even more in the differences in the response to these therapies in different patient subpopulations. The purpose of this study is to assess the demographic and clinical charateristics, treatment patterns and incidence of events (discontinuation, persistence, key primary clinical outcomes) in NVAF patients that initiated OACs in study period.

#### 6. RESEARCH QUESTION AND OBJECTIVES

## Primary Objectives

- To assess demographic and clinical characteristics of NVAF patients treated with oral anticoagulants (OACs) in Colombia.
- To describe treatment patterns (eg. OAC usage, dose, concomitant medications, persistence)

#### **Exploratory Objectives**

• To descriptively assess the time to clinical events (Effectiveness and Safety Outcomes) among patients persistent on OAC therapy.

Effectiveness outcomes: First Stroke/ Systemic Embolism;

Safety outcomes: Major bleeding, CCI

#### 7. RESEARCH METHODS

#### 7.1. Study Design

Observational, descriptive study of a retrospective cohort of adult patients diagnosed with NVAF in selected Health Maintenance Organization (HMO) of Colombia. These patients will be identified from the drug claim database, whose index date of the study will be the first prescription with any of the oral anticoagulants, that is, they are patients with NVAF for the first time starting a therapy with any of the NOACs between January 1, 2013 and June 30, 2018 and follow up period will be among January 2013 to July 2019, to ensure that the last patients can provide follow-up for one year. Patients will be required to have an NVAF diagnosis before or on the index date and health plan for 6 months pre-index date (baseline period).

Following, it will be verified that the patients meet the inclusion and exclusion criteria of the study. Once patients are selected and with the index date of each patient, they will be followed-up until discontinuation, switch of treatment, death or first event of stroke/ systemic embolism, major bleeding event, death or end of follow-up. Patients who are lost to follow-up, change of HMO and do not have access to the medical record will be considered as missing (Figure 1).



Figure 1. Study Design

The information will be analyzed in two moments: (i) the period of the index date, where the baseline information of patients will be collected; (ii) and the follow-up period, during this period the clinical results will be evaluated as well as the continuation of the treatment in the study population and for specific subpopulations.

Those patients who initiated treatment with any oral anticoagulant between January 2013 and June 30, 2018 will be included. This means that patients who start warfarin and NOACs would

be included within this period. Patients who initiate NOACs within the established period and who have been exposed to warfarin before 2013 will also be included.

Only the exposure period will be considered with the initial treatment, even in those patients who were on warfarin treatment before 2013, in the latter, the follow-up will be the treatment initiation with a NOAC in case of change after 2013. Follow-up will be carried out until the patient has a switch of treatment, discontinuation, death, first stroke/ systemic embolism, or major bleeding, or until end of follow-up, June 30, 2019 (Figure 2).



Figure 2. Inclusion of Patients

#### 7.2. Setting

The study will be conducted with the Audifarma patient cohort that meets the inclusion and exclusion criteria between the periods from January 2013 to June 30, 2018. The follow up period will be among January 2013 to July 2019, to ensure that the last patients can provide follow-up for one year.

This study will include the entire population in which medical records can be accessed. This will depend on the authorization of the HMOs for review of medical records. Participating patients will be followed-up until the patient has a stroke/systemic embolism, major bleeding, discontinuation, change of treatment or until the data collection period is completed.

#### 7.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- Patients with a diagnosis of AF considered according to the following diagnoses as per the ICD I48 codes at some point before or on the index date, without recorded valvular disease;
- b) Patients who have started treatment with apixaban, dabigatran, rivaroxaban and warfarin for the first time during the identification period, understanding as start of drug delivery by insurer, and after the diagnosis of AF between January 1, 2013 to June 30, 2018;
- c) Patients starting apixaban, dabigatran, rivaroxaban from January 1, 2013 to June 30, 2018 in patients previously exposed to warfarin;
- d) Patient had continuous health plan for 6 months pre-index date (baseline period);
- e) Patients older than 18 years old on the index date;
- f) NVAF diagnosis before or on the index date

#### 7.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

- e) Patients with any of the following diagnoses prior to the use of the treatments of interest or index date:
  - Valvular heart disease or valve replacement ICD-10 codes: I05, I06, I07, I08, I09, I22, I34, I35, I36, I37, I38, I39, I700, I702-I709; Q22, Q23, Q25, T82,Z95.
  - Pregnancy during the study period. ICD-10 O00-O9A
  - Diagnosis of venous thromboembolism (VTE) ICD-10 codes: I26, I80 I82;
- f) Individuals with a transitory diagnosis of NVAF prior to the use of the treatments of interest or index date;
- g) Exposure to more than one OAC on or after the index date, during the follow-up period.
- h) NOAC doses different from those recommended by the manufacturing laboratories.

#### **7.2.3.** Cohorts

After applying the inclusion and exclusion criteria, eligible patients will be assigned to the following four cohorts based on the OAC received on the index date.

1. Apixaban

- 2. Dabigatran
- 3. Rivaroxaban
- 4. Warfarin

Depending on the dosage of the NOAC prescribed on the index date, and in comparison to the standard conventions of total daily doses, patients may be classified into 3 different groups:

- **High doses:** apixaban 10 mg/day rivaroxaban: 20 mg/day dabigatran: 300 mg/day;
- Low doses: apixaban 5 mg/day rivaroxaban: 15 mg/day dabigatran: 220 mg/day
- Other doses: to be excluded, doses not recommended by the manufacturing laboratories.

#### 7.3. Variables

The described variables are classified into two variable groups according to the role, the clinical outcome and baseline (demographic, clinical, treatment variables). The latter include the possible subgroups to consider. These analyses are initially exploratory to the extent that the specific analyses may be performed according to the sample collected.

**Table 1. Table of Variables** 

| Variable | Role | Data source (s) | Operational definition |
|---|---|---|---|
| Age | Demographic characteristic | Medical record | Birthday |
| Gender | Demographic characteristic | Medical record | Male, female, other |
| Race | Demographic characteristic | Medical record | White, half-breed, indigenous, black, others |
| Weight | Demographic characteristic | Medical record | Kg |
| Height | Demographic characteristic | Medical record | Mt (meters) |
| Body mass index | Demographic characteristic | Medical record | Kg/mt2 |
| City of residence | Demographic characteristic | Medical record | Cities of Colombia |
| Time to diagnosis to NVAF | Clinical characteristic | Medical record | Date (dd/mm/yy) |
| High alcohol intake at OAC prescription date | Clinical characteristic | Medical record | Yes, No |

| Variable | Role | Data source (s) | Operational definition |
|---|---|---|---|
| Diabetes | Clinical characteristic | Medical record | No, without chronic complication, with end-organ damage |
| Liver disease | Clinical characteristic | Medical record | No, mild,<br>moderade, severe |
| Hypertension | Clinical characteristic | Medical record | Diagnosis of hypertension (Yes, No) |
| Uncontrolled hypertension at OAC prescription date | Clinical characteristic | Medical record | Yes, No |
| Rheumatic disease | Clinical characteristic | Medical record | Yes, No |
| Acquired Immune<br>Deficiency Syndrome<br>(AIDS) | Clinical characteristic | Medical record | Yes, No |
| Severe renal disease<br>(dialysis, organ<br>transplant) | Clinical characteristic | Medical record | Yes, No |
| Moderade renal<br>disease (creatinine ><br>3 mg/dL) | Clinical characteristic | Medical record | Yes, No |
| Chronic heart failure | Clinical characteristic | Medical record | Yes, No |
| Myocardial infarction | Clinical characteristic | Medical record | Yes, No |
| Chronic obstructive pulmonary disease (COPD) | Clinical characteristic | Medical record | Yes, No |
| Peripheral vascular disease | Clinical characteristic | Medical record | Yes, No |
| Stroke or transient ischemic attack (TIA) | Clinical characteristic | Medical record | Yes, No |
| Dementia | Clinical characteristic | Medical record | Yes, No |
| Hemiplegia | Clinical characteristic | Medical record | Yes, No |
| Connective tissue disease | Clinical characteristic | Medical record | Yes, No |
| Leukemia | Clinical characteristic | Medical record | Yes, No |

| Variable | Role | Data source (s) | Operational definition |
|---|---|---|---|
| Malignant lymphoma | Clinical characteristic | Medical record | Yes, No |
| Peptic ulcer disease | Clinical characteristic | Medical record | Yes, No |
| Metastatic solid tumor | Clinical characteristic | Medical record | Yes, No |
| History of ischemic<br>or hemorrhagic<br>stroke | Clinical characteristic | Medical record | Yes, No |
| History of TIA | Clinical characteristic | Medical record | Yes, No |
| History of de tromboembolismo | Clinical characteristic | Medical record | Yes, No |
| Enfermedad coronaria | Clinical characteristic | Medical record | Yes, No |
| History of de<br>hemorragia<br>gastrointestinal | Clinical characteristic | Medical record | Yes, No |
| History of Intracranial bleeding | Clinical characteristic | Medical record | Yes, No |
| History of Other bleeding | Clinical characteristic | Medical record | Yes, No |
| Bleeding history or predisposition at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| INR > 60% at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| Use of aspirin at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| Use of clopidogrel at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| Use of NSAIDs at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| HASBLED at start OAC treatment | Clinical characteristic | Medical record | Score – number higher than 0 |
| CHA2DS2-VASc at start OAC treatment | Clinical characteristic | Medical record | Score – number higher than 0 |
| Anaemia at start OAC treatment | Clinical characteristic | Medical record | Yes, No |
| Stroke Time to stroke | Clinical outcome Clinical outcome | Medical record Medical record | Yes, No Date of event dd/mm/yy |

| Variable | Role | Data source (s) | Operational definition |
|---|---|---|---|
| Type of stroke | Clinical outcome | Medical record | Ischemic stroke,<br>Haemorrhagic or<br>not specified |
| Pulmonary embolism | Clinical outcome | Medical record | Yes, No |
| Time to pulmonary embolism | Clinical outcome | Medical record | Date of event dd/mm/yy |
| Gastrointestinal bleeding | Clinical outcome | Medical record | Yes, No |
| Time to gastrointestinal bleeding | Clinical outcome | Medical record | Date of event dd/mm/yy |
| Intracranial bleeding | Clinical outcome | Medical record | Yes, No |
| Time to Intracranial bleeding | Clinical outcome | Medical record | Date of event dd/mm/yy |
| Other major bleeding | Clinical outcome | Medical record | Yes, No |
| Time to other major bleeding | Clinical outcome | Medical record | Date of event dd/mm/yy |
| | | | V. N |
| Persistence | Clinical outcome | Claim databases | Yes, No |
| OAC treatment | Treatment | Claim databases | Warfarin, apixaban,<br>rivaroxaban,<br>dabigatran |
| Diagnosis at index date | Treatment | Claim databases | Diagnosis AF based<br>on ICD-10 |
| Date of OAC prescription | Treatment | Claim databases | Date reported dd/mm/yy |
| Dosage of the initial OAC treatment | Treatment | Claim databases | Mg per dose |
| Initial frequency of OAC treatment | Treatment | Claim databases | Number of doses at initial OAC treatment |
| OAC escalation | Treatment | Claim databases | Yes, No |
| Type of OAC escalation | Treatment | Claim databases | Dose increase or dose decrease |
| Time to OAC escalation | Treatment | Claim databases | Date reported dd/mm/yy |
| CCI | | | |

| Variable | Role | Data source (s) | Operational definition |
|---|---|---|---|
| CCI | | | |
| INR testing monthly in patients with warfarin | Treatment | Medical record | INR reported in the medical record per month |
| Switch to another OAC treatment: | Treatment | Claim databases | Yes, No |
| Time to Switch to another OAC treatment | Treatment | Claim databases | Date reported dd/mm/yy |
| Causa de cambio | Treatment | Medical record | Adverse events, effectiveness, adherence, patient preference, administrative problems, not reported, others |
| Concomitant therapies by OAC prescription | Treatment | Medical record | NSAIDs, Angiotensin-converting- enzyme (ACE) inhibitors, Amiodarone, Beta- blockers, Angiotensin II receptor blockers (ARBs), Aspirin, Clopidogrel, Digoxin, Diuretics, calcium blockers, statins, proton pump inhibitor, selective H2 antagonists, antidiabetics, insulin, serotonin reuptake inhibitors |
| Previously exposed to warfarin | Treatment | Claim databases | Yes, No |

#### 7.3.1. Definition of outcome variables

• OAC escalation: The dose escalation of the OAC dose will be considered as a dose frequency according to the index dose, as well as the follow-up doses. The proportion of patients experiencing "dose increase", "dose decrease" or "no change" during follow-up with respect to the index dose will be measured, and the time to dose increase or decrease will be calculated.



- **Switch of treatment:** A switch among anticoagulants will be defined as a prescription filled for non-index anticoagulants within +/- 30 days after the date of discontinuation.
- **Persistence:** Persistence will be defined as the time under OAC therapy, calculated as the time in days from the index date to the date of discontinuation or change to treatment. As previously stated, discontinuation will be defined as a change of treatment, that is, to another OAC, or when there is no evidence of a prescription for 60 days from the last supply delivered, whichever comes first.

Therefore, if a patient does not receive his next prescription for the OAC therapy within 60 days after the end of the previous prescription, it will be considered that he discontinued therapy, and the date of the last prescription will be considered as the final date of persistence.

Persistence with OAC therapy will be considered during the period of individual patient follow-up. Patients will be censored at the end of their follow-up period.

• **Major bleeding:** Patients presenting any of the following diagnoses during the follow-up period:

| ICD-10 | Description |
|--------|---------------------------------------------------------|
| I60 | Subarachnoid haemorrhage |
| I61 | Intracerebral haemorrhage |
| I62 | Other nontraumatic intracranial haemorrhage |
| I690 | Sequelae of subarachnoid haemorrhage |
| I691 | Sequelae of intracerebral haemorrhage |
| I692 | Sequelae of other nontraumatic intracranial haemorrhage |
| S064 | Epidural haemorrhage |
| S065 | Traumatic subdural haemorrhage |
| S066 | Traumatic subarachnoid haemorrhage |
| I850 | Oesophageal varices with bleeding |
| K250 | Acute with haemorrhage |

| ICD-10 | Description |
|--------|--------------------------------------------------------------|
| K252 | Acute with both haemorrhage and perforation |
| K254 | Chronic or unspecified with haemorrhage |
| K256 | Chronic or unspecified with both haemorrhage and perforation |
| K260 | Acute with haemorrhage |
| K262 | Acute with both haemorrhage and perforation |
| K264 | Chronic or unspecified with haemorrhage |
| K266 | Chronic or unspecified with both haemorrhage and perforation |
| K270 | Acute with haemorrhage |
| K272 | Acute with both haemorrhage and perforation |
| K274 | Chronic or unspecified with haemorrhage |
| K276 | Chronic or unspecified with both haemorrhage and perforation |
| K280 | Acute with haemorrhage |
| K282 | Acute with both haemorrhage and perforation |
| K284 | Chronic or unspecified with haemorrhage |
| K286 | Chronic or unspecified with both haemorrhage and perforation |
| K290 | Acute haemorrhagic gastritis |
| K625 | Haemorrhage of anus and rectum |
| K920 | Haematemesis |
| K921 | Melaena |
| K922 | Gastro-intestinal haemorrhage, unspecified |
| D62 | Acute posthaemorrhagic anaemia |
| H356 | Retinal haemorrhage |
| H431 | Vitreous haemorrhage |
| H450 | Vitreous haemorrhage in diseases classified elsewhere |
| H922 | Otorrhagia |
| I312 | Haemopericardium, not elsewhere classified |
| J942 | Haemothorax |
| R04 | Haemorrhage from respiratory passages |
| K661 | Haemoperitoneum |
| M250 | Haemarthrosis |
| N02 | Recurrent and persistent haematuria |
| N938 | Other specified abnormal uterine and vaginal bleeding |
| N939 | Abnormal uterine and vaginal bleeding, unspecified |
| N950 | Postmenopausal bleeding |
| R31 | Unspecified haematuria |
| R58 | Haemorrhage, not elsewhere classified |
| T792 | Traumatic secondary and recurrent haemorrhage |

• **Ischemic stroke:** Patients who report the following diagnoses in the medical history during the follow-up period:

| ICD-10 | Description |
|--------|----------------------------------------------------|
| I63 | Cerebral infarction |
| I64 | Stroke, not specified as haemorrhage or infarction |

Except I63.6 Cerebral infarction due to thrombosis of cerebral veins, non-pyogenic

• **Hemorrhagic stroke:** Patients presenting the following diagnosis in the medical record:

| ICD-10 | Description |
|--------|---------------------------------------------|
| I60 | Subarachnoid haemorrhage |
| I61 | Intracerebral haemorrhage |
| I62 | Other nontraumatic intracranial haemorrhage |

• Systemic embolism: Patients who report any of the following diagnoses:

| ICD-10 | Description |
|--------|----------------------------------|
| I74 | Arterial embolism and thrombosis |

#### Definition of covariates

• Age: Categorical variable, continues in years. It will be defined from the index date and will be used to assign patients to the following age categories:

18 - 49

50 - 59

60 - 69

70 - 79

 $\geq$  80 years old.

• **Charlson Index**: Charlson comorbidity index will be created during the reference period taking into account the following score:

#### 1 point each:

Myocardial infarction

| ICD-10 | Description |
|--------|----------------------------------|
| I21 | Acute myocardial infarction |
| I22 | Subsequent myocardial infarction |
| I252 | Old myocardial infarction |

#### • Congestive heart failure

| ICD-10 | Description |
|---|---|
| I110 | Hypertensive heart disease with (congestive) heart failure |
| I130 | Hypertensive heart and renal disease with (congestive) heart failure |
| I132 | Hypertensive heart and renal disease with both (congestive) heart failure and renal failure |
| I110 | Hypertensive heart disease with (congestive) heart failure |

#### Peripheral vascular disease

| ICD-10 | Description |
|--------|----------------------------------------------|
| I70 | Atherosclerosis |
| I71 | Aortic aneurysm and dissection |
| I731 | Thromboangiitis obliterans [Buerger] |
| I738 | Other specified peripheral vascular diseases |
| I739 | Peripheral vascular disease, unspecified |

| ICD-10 | Description |
|--------|-----------------------------------------------------------------|
| I771 | Stricture of artery |
| I790 | Aneurysm of aorta in diseases classified elsewhere |
| I792 | Peripheral angiopathy in diseases classified elsewhere |
| K551 | Chronic vascular disorders of intestine |
| K558 | Other vascular disorders of intestine |
| K559 | Vascular disorder of intestine, unspecified |
| Z958 | Presence of other cardiac and vascular implants and grafts |
| Z959 | Presence of cardiac and vascular implant and graft, unspecified |

#### Dementia

| ICD-10 | Description |
|--------|--------------------------------------------------------|
| F00 | Dementia in Alzheimer's disease |
| F01 | Vascular dementia |
| F02 | Dementia in other diseases classified elsewhere |
| F03 | Unspecified dementia |
| G30 | Alzheimer's disease |
| F051 | Delirium superimposed on dementia |
| G311 | Senile degeneration of brain, not elsewhere classified |

### Cerebrovascular disease

| ICD-10 | Description |
|---|---|
| G45 | Transient cerebral ischaemic attacks and related syndromes |
| G46 | Vascular syndromes of brain in cerebrovascular diseases |
| I60 | Subarachnoid haemorrhage |
| I61 | Intracerebral haemorrhage |
| I62 | Other nontraumatic intracranial haemorrhage |
| I63 | Cerebral infarction |
| I64 | Stroke, not specified as haemorrhage or infarction |
| I65 | Occlusion and stenosis of precerebral arteries, not resulting in cerebral infarction |
| I66 | Occlusion and stenosis of cerebral arteries, not resulting in cerebral infarction |
| I67 | Other cerebrovascular diseases |
| I68 | Cerebrovascular disorders in diseases classified elsewhere |
| I69 | Sequelae of cerebrovascular disease |
| H340 | Transient retinal artery occlusion |

#### Chronic pulmonary disease

| ICD-10 | Description |
|--------|---------------------------------------------------------|
| J40 | Bronchitis, not specified as acute or chronic |
| J41 | Simple and mucopurulent chronic bronchitis |
| J42 | Unspecified chronic bronchitis |
| J43 | Emphysema |
| J44 | Other chronic obstructive pulmonary disease |
| J45 | Asthma |
| J46 | Status asthmaticus |
| J47 | Bronchiectasis |
| J60 | Coalworker's pneumoconiosis |
| J61 | Pneumoconiosis due to asbestos and other mineral fibres |
| J62 | Pneumoconiosis due to dust containing silica |

## Apixaban B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

#### Final, 10 October 2019

| ICD-10 | Description |
|---|---|
| J63 | Pneumoconiosis due to other inorganic dusts |
| J64 | Unspecified pneumoconiosis |
| J65 | Pneumoconiosis associated with tuberculosis |
| J66 | Airway disease due to specific organic dust |
| J67 | Hypersensitivity pneumonitis due to organic dust |
| I278 | Other specified pulmonary heart diseases |
| I279 | Pulmonary heart disease, unspecified |
| J684 | Chronic respiratory conditions due to chemicals, gases, fumes and vapours |
| J701 | Chronic and other pulmonary manifestations due to radiation |
| J703 | Chronic drug-induced interstitial lung disorders |

#### Connective tissue disease

| ICD-10 | Description |
|--------|--------------------------------------------------|
| M05 | Seropositive rheumatoid arthritis |
| M06 | Other rheumatoid arthritis |
| M32 | Systemic lupus erythematosus |
| M33 | Dermatopolymyositis |
| M34 | Systemic sclerosis |
| M315 | Giant cell arteritis with polymyalgia rheumatica |
| M351 | Other overlap syndromes |
| M353 | Polymyalgia rheumatica |
| M360 | Dermato(poly)myositis in neoplastic disease |

#### Ulcer disease

| ICD-10 | Description |
|--------|--------------------------------|
| K25 | Gastric ulcer |
| K26 | Duodenal ulcer |
| K27 | Peptic ulcer, site unspecified |
| K28 | Gastrojejunal ulcer |

#### Mild liver disease

| ICD-10 | Description |
|--------|----------------------------------------------------------|
| B18 | Chronic viral hepatitis |
| K73 | Chronic hepatitis, not elsewhere classified |
| K74 | Fibrosis and cirrhosis of liver |
| K700 | Alcoholic fatty liver |
| K701 | Alcoholic hepatitis |
| K702 | Alcoholic fibrosis and sclerosis of liver |
| K703 | Alcoholic cirrhosis of liver |
| K709 | Alcoholic liver disease, unspecified |
| K717 | Toxic liver disease with fibrosis and cirrhosis of liver |
| K713 | Toxic liver disease with chronic persistent hepatitis |
| K714 | Toxic liver disease with chronic lobular hepatitis |
| K715 | Toxic liver disease with chronic active hepatitis |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K762 | Central haemorrhagic necrosis of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K768 | Other specified diseases of liver |
| K769 | Liver disease, unspecified |
| Z944 | Liver transplant status |
| B18 | Chronic viral hepatitis |
| K73 | Chronic hepatitis, not elsewhere classified |
| K74 | Fibrosis and cirrhosis of liver |
| K700 | Alcoholic fatty liver |
| K701 | Alcoholic hepatitis |
| K702 | Alcoholic fibrosis and sclerosis of liver |
| K703 | Alcoholic cirrhosis of liver |
| K709 | Alcoholic liver disease, unspecified |
| K717 | Toxic liver disease with fibrosis and cirrhosis of liver |
| K713 | Toxic liver disease with chronic persistent hepatitis |
| K714 | Toxic liver disease with chronic lobular hepatitis |

## Apixaban B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

#### Final, 10 October 2019

| ICD-10 | Description |
|--------|---------------------------------------------------|
| K715 | Toxic liver disease with chronic active hepatitis |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K762 | Central haemorrhagic necrosis of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K768 | Other specified diseases of liver |
| K769 | Liver disease, unspecified |
| Z944 | Liver transplant status |

### • Diabetes without chronic complication

| ICD-10 | Description |
|---|---|
| E100 | Insulin-dependent diabetes mellitus with coma |
| E101 | Insulin-dependent diabetes mellitus with ketoacidosis |
| E106 | Insulin-dependent diabetes mellitus with other specified complications |
| E108 | Insulin-dependent diabetes mellitus with unspecified complications |
| E109 | Insulin-dependent diabetes mellitus without complications |
| E110 | Non-insulin-dependent diabetes mellitus with coma |
| E111 | Non-insulin-dependent diabetes mellitus with ketoacidosis |
| E116 | Non-insulin-dependent diabetes mellitus with other specified complications |
| E118 | Non-insulin-dependent diabetes mellitus with unspecified complications |
| E119 | Non-insulin-dependent diabetes mellitus without complications |
| E120 | Malnutrition-related diabetes mellitus with coma |
| E121 | Malnutrition-related diabetes mellitus with ketoacidosis |
| E126 | Malnutrition-related diabetes mellitus with other specified complications |
| E128 | Malnutrition-related diabetes mellitus with unspecified complications |
| E129 | Malnutrition-related diabetes mellitus without complications |
| E130 | Other specified diabetes mellitus with coma |
| E131 | Other specified diabetes mellitus with ketoacidosis |
| E136 | Other specified diabetes mellitus with other specified complications |
| E138 | Other specified diabetes mellitus with unspecified complications |
| E139 | Other specified diabetes mellitus without complications |
| E140 | Unspecified diabetes mellitus with coma |
| E141 | Unspecified diabetes mellitus with ketoacidosis |
| E146 | Unspecified diabetes mellitus with other specified complications |
| E148 | Unspecified diabetes mellitus with unspecified complications |
| E149 | Unspecified diabetes mellitus without complications |
| E100 | Insulin-dependent diabetes mellitus with coma |
| E101 | Insulin-dependent diabetes mellitus with ketoacidosis |
| E106 | Insulin-dependent diabetes mellitus with other specified complications |
| E108 | Insulin-dependent diabetes mellitus with unspecified complications |
| E109 | Insulin-dependent diabetes mellitus without complications |
| E110 | Non-insulin-dependent diabetes mellitus with coma |
| E111 | Non-insulin-dependent diabetes mellitus with ketoacidosis |
| E116 | Non-insulin-dependent diabetes mellitus with other specified complications |
| E118 | Non-insulin-dependent diabetes mellitus with unspecified complications |
| E119 | Non-insulin-dependent diabetes mellitus without complications |
| E120 | Malnutrition-related diabetes mellitus with coma |
| E121 | Malnutrition-related diabetes mellitus with ketoacidosis |
| E126 | Malnutrition-related diabetes mellitus with other specified complications |
| E128 | Malnutrition-related diabetes mellitus with unspecified complications |
| E129 | Malnutrition-related diabetes mellitus without complications |

| ICD-10 | Description |
|---|---|
| E130 | Other specified diabetes mellitus with coma |
| E131 | Other specified diabetes mellitus with ketoacidosis |
| E136 | Other specified diabetes mellitus with other specified complications |
| E138 | Other specified diabetes mellitus with unspecified complications |
| E139 | Other specified diabetes mellitus without complications |
| E140 | Unspecified diabetes mellitus with coma |
| E141 | Unspecified diabetes mellitus with ketoacidosis |
| E146 | Unspecified diabetes mellitus with other specified complications |
| E148 | Unspecified diabetes mellitus with unspecified complications |
| E149 | Unspecified diabetes mellitus without complications |

#### 2 point each:

### Hemiplegia or paraplegia

| ICD-10 | Description |
|--------|---------------------------------|
| G81 | Hemiplegia |
| G82 | Paraplegia and tetraplegia |
| G041 | Tropical spastic paraplegia |
| G114 | Hereditary spastic paraplegia |
| G801 | Spastic diplegia |
| G802 | Infantile hemiplegia |
| G830 | Diplegia of upper limbs |
| G831 | Monoplegia of lower limb |
| G832 | Monoplegia of upper limb |
| G833 | Monoplegia, unspecified |
| G834 | Cauda equina syndrome |
| G839 | Paralytic syndrome, unspecified |
| G81 | Hemiplegia |
| G82 | Paraplegia and tetraplegia |
| G041 | Tropical spastic paraplegia |
| G114 | Hereditary spastic paraplegia |
| G801 | Spastic diplegia |
| G802 | Infantile hemiplegia |
| G830 | Diplegia of upper limbs |
| G831 | Monoplegia of lower limb |
| G832 | Monoplegia of upper limb |
| G833 | Monoplegia, unspecified |
| G834 | Cauda equina syndrome |
| G839 | Paralytic syndrome, unspecified |

#### ■ *Moderate or severe renal disease*

| ICD-10 | Description |
|--------|--------------------------------------------------------|
| N18 | Chronic renal failure |
| N19 | Unspecified renal failure |
| N052 | Diffuse membranous glomerulonephritis |
| N053 | Diffuse mesangial proliferative glomerulonephritis |
| N054 | Diffuse endocapillary proliferative glomerulonephritis |
| N055 | Diffuse mesangiocapillary glomerulonephritis |
| N056 | Dense deposit disease |
| N057 | Diffuse crescentic glomerulonephritis |

| ICD-10 | Description |
|--------|---------------------------------------------------------|
| N250 | Renal osteodystrophy |
| I120 | Hypertensive renal disease with renal failure |
| I131 | Hypertensive heart and renal disease with renal failure |
| N032 | Diffuse membranous glomerulonephritis |
| N033 | Diffuse mesangial proliferative glomerulonephritis |
| N034 | Diffuse endocapillary proliferative glomerulonephritis |
| N035 | Diffuse mesangiocapillary glomerulonephritis |
| N036 | Dense deposit disease |
| N037 | Diffuse crescentic glomerulonephritis |
| Z490 | Preparatory care for dialysis |
| Z491 | Extracorporeal dialysis |
| Z492 | Other dialysis |
| Z940 | Kidney transplant status |
| Z992 | Dependence on renal dialysis |

### Diabetes with end-organ damage

| ICD-10 | Description |
|---|---|
| E102 | Insulin-dependent diabetes mellitus with renal complications |
| E103 | Insulin-dependent diabetes mellitus with ophthalmic complications |
| E104 | Insulin-dependent diabetes mellitus with neurological complications |
| E105 | Insulin-dependent diabetes mellitus with peripheral circulatory complications |
| E107 | Insulin-dependent diabetes mellitus with multiple complications |
| E112 | Non-insulin-dependent diabetes mellitus with renal complications |
| E113 | Non-insulin-dependent diabetes mellitus with ophthalmic complications |
| E114 | Non-insulin-dependent diabetes mellitus with neurological complications |
| E115 | Non-insulin-dependent diabetes mellitus with peripheral circulatory complications |
| E117 | Non-insulin-dependent diabetes mellitus with multiple complications |
| E122 | Malnutrition-related diabetes mellitus with renal complications |
| E123 | Malnutrition-related diabetes mellitus with ophthalmic complications |
| E124 | Malnutrition-related diabetes mellitus with neurological complications |
| E125 | Malnutrition-related diabetes mellitus with peripheral circulatory complications |
| E127 | Malnutrition-related diabetes mellitus with multiple complications |
| E132 | Other specified diabetes mellitus with renal complications |
| E133 | Other specified diabetes mellitus with ophthalmic complications |
| E134 | Other specified diabetes mellitus with neurological complications |
| E135 | Other specified diabetes mellitus with peripheral circulatory complications |
| E137 | Other specified diabetes mellitus with multiple complications |
| E142 | Unspecified diabetes mellitus with renal complications |
| E143 | Unspecified diabetes mellitus with ophthalmic complications |
| E144 | Unspecified diabetes mellitus with neurological complications |
| E145 | Unspecified diabetes mellitus with peripheral circulatory complications |
| E147 | Unspecified diabetes mellitus with multiple complications |
| E102 | Insulin-dependent diabetes mellitus with renal complications |
| E103 | Insulin-dependent diabetes mellitus with ophthalmic complications |
| E104 | Insulin-dependent diabetes mellitus with neurological complications |
| E105 | Insulin-dependent diabetes mellitus with peripheral circulatory complications |
| E107 | Insulin-dependent diabetes mellitus with multiple complications |
| E112 | Non-insulin-dependent diabetes mellitus with renal complications |
| E113 | Non-insulin-dependent diabetes mellitus with ophthalmic complications |
| E114 | Non-insulin-dependent diabetes mellitus with neurological complications |
| E115 | Non-insulin-dependent diabetes mellitus with peripheral circulatory complications |

## Apixaban B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

#### Final, 10 October 2019

| ICD-10 | Description |
|---|---|
| E117 | Non-insulin-dependent diabetes mellitus with multiple complications |
| E122 | Malnutrition-related diabetes mellitus with renal complications |
| E123 | Malnutrition-related diabetes mellitus with ophthalmic complications |
| E124 | Malnutrition-related diabetes mellitus with neurological complications |
| E125 | Malnutrition-related diabetes mellitus with peripheral circulatory complications |
| E127 | Malnutrition-related diabetes mellitus with multiple complications |
| E132 | Other specified diabetes mellitus with renal complications |
| E133 | Other specified diabetes mellitus with ophthalmic complications |
| E134 | Other specified diabetes mellitus with neurological complications |
| E135 | Other specified diabetes mellitus with peripheral circulatory complications |
| E137 | Other specified diabetes mellitus with multiple complications |
| E142 | Unspecified diabetes mellitus with renal complications |
| E143 | Unspecified diabetes mellitus with ophthalmic complications |
| E144 | Unspecified diabetes mellitus with neurological complications |
| E145 | Unspecified diabetes mellitus with peripheral circulatory complications |
| E147 | Unspecified diabetes mellitus with multiple complications |

Any tumor (including lymphoma and leukemia except malignant neoplasms of

| | SKIN) |
|---|---|
| ICD-<br>10 | Description |
| C00 | Malignant neoplasm of lip |
| C01 | Malignant neoplasm of base of tongue |
| C02 | Malignant neoplasm of other and unspecified parts of tongue |
| C03 | Malignant neoplasm of gum |
| C04 | Malignant neoplasm of floor of mouth |
| C05 | Malignant neoplasm of palate |
| C06 | Malignant neoplasm of other and unspecified parts of mouth |
| C07 | Malignant neoplasm of parotid gland |
| C08 | Malignant neoplasm of other and unspecified major salivary glands |
| C09 | Malignant neoplasm of tonsil |
| C10 | Malignant neoplasm of oropharynx |
| C11 | Malignant neoplasm of nasopharynx |
| C12 | Malignant neoplasm of pyriform sinus |
| C13 | Malignant neoplasm of hypopharynx |
| C14 | Malignant neoplasm of other and ill-defined sites in the lip, oral cavity and pharynx |
| C15 | Malignant neoplasm of oesophagus |
| C16 | Malignant neoplasm of stomach |
| C17 | Malignant neoplasm of small intestine |
| C18 | Malignant neoplasm of colon |
| C19 | Malignant neoplasm of rectosigmoid junction |
| C20 | Malignant neoplasm of rectum |
| C21 | Malignant neoplasm of anus and anal canal |
| C22 | Malignant neoplasm of liver and intrahepatic bile ducts |
| C23 | Malignant neoplasm of gallbladder |
| C24 | Malignant neoplasm of other and unspecified parts of biliary tract |
| C25 | Malignant neoplasm of pancreas |
| C26 | Malignant neoplasm of other and ill-defined digestive organs |
| C30 | Malignant neoplasm of nasal cavity and middle ear |
| C31 | Malignant neoplasm of accessory sinuses |
| C32 | Malignant neoplasm of larynx |
| C33 | Malignant neoplasm of trachea |
| C34 | Malignant neoplasm of bronchus and lung |
| C37 | Malignant neoplasm of thymus |
| C38 | Malignant neoplasm of heart, mediastinum and pleura |
| C39 | Malignant neoplasm of other and ill-defined sites in the respiratory system and intrathoracic organs |
| C40 | Malignant neoplasm of bone and articular cartilage of limbs |
| C41 | Malignant neoplasm of bone and articular cartilage of other and unspecified sites |
| C43 | Malignant melanoma of skin |
| C45 | Mesothelioma |
| C46 | Kaposi's sarcoma |
| C47 | Malignant neoplasm of peripheral nerves and autonomic nervous system |
| C48 | Malignant neoplasm of retroperitoneum and peritoneum |
| C49 | Malignant neoplasm of other connective and soft tissue |
| C50 | Malignant neoplasm of breast |
| C51 | Malignant neoplasm of vulva |
| C52 | Malignant neoplasm of vagina |
| C53 | Malignant neoplasm of cervix uteri |

## Apixaban B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

#### Final, 10 October 2019

| ICD-<br>10 | Description |
|---|---|
| C54 | Malignant neoplasm of corpus uteri |
| C55 | Malignant neoplasm of uterus, part unspecified |
| C56 | Malignant neoplasm of ovary |
| C57 | Malignant neoplasm of other and unspecified female genital organs |
| C58 | Malignant neoplasm of placenta |
| C60 | Malignant neoplasm of penis |
| C61 | Malignant neoplasm of prostate |
| C62 | Malignant neoplasm of testis |
| C63 | Malignant neoplasm of other and unspecified male genital organs |
| C64 | Malignant neoplasm of kidney, except renal pelvis |
| C65 | Malignant neoplasm of renal pelvis |
| C66 | Malignant neoplasm of ureter |
| C67 | Malignant neoplasm of bladder |
| C68 | Malignant neoplasm of other and unspecified urinary organs |
| C69 | Malignant neoplasm of eye and adnexa |
| C70 | Malignant neoplasm of meninges |
| C71 | Malignant neoplasm of brain |
| C72 | Malignant neoplasm of spinal cord, cranial nerves and other parts of central nervous system |
| C73 | Malignant neoplasm of thyroid gland |
| C74 | Malignant neoplasm of adrenal gland |
| C75 | Malignant neoplasm of other endocrine glands and related structures |
| C76 | Malignant neoplasm of other and ill-defined sites |
| C81 | Hodgkin's disease |
| C82 | Follicular [nodular] non-Hodgkin's lymphoma |
| C83 | Diffuse non-Hodgkin's lymphoma |
| C84 | Peripheral and cutaneous T-cell lymphomas |
| C85 | Other and unspecified types of non-Hodgkin's lymphoma |
| C88 | Malignant immunoproliferative diseases |
| C90 | Multiple myeloma and malignant plasma cell neoplasms |
| C91 | Lymphoid leukaemia |
| C92 | Myeloid leukaemia |
| C93 | Monocytic leukaemia |
| C94 | Other leukaemias of specified cell type |
| C95 | Leukaemia of unspecified cell type |
| C96 | Other and unspecified malignant neoplasms of lymphoid, haematopoietic and related tissue |
| C97 | Malignant neoplasms of independent (primary) multiple sites |

#### 3 points each:

Moderate or severe liver disease

| ICD-10 | Description |
|--------|------------------------------------------------------|
| K704 | Alcoholic hepatic failure |
| K711 | Toxic liver disease with hepatic necrosis |
| K721 | Chronic hepatic failure |
| K729 | Hepatic failure, unspecified |
| K765 | Hepatic veno-occlusive disease |
| K766 | Portal hypertension |
| K767 | Hepatorenal syndrome |
| I850 | Oesophageal varices with bleeding |
| I859 | Oesophageal varices without bleeding |
| I864 | Gastric varices |
| 1982 | Oesophageal varices in diseases classified elsewhere |

#### 6 points each:

• *Metastatic solid tumor* 

| ICD-10 | Description |
|--------|------------------------------------------------------------------|
| C77 | Secondary and unspecified malignant neoplasm of lymph nodes |
| C78 | Secondary malignant neoplasm of respiratory and digestive organs |
| C79 | Secondary malignant neoplasm of other sites |
| C80 | Malignant neoplasm without specification of site |

■ Human immunodeficiency virus (HIV)-AIDS

| ICD-10 | Description |
|---|---|
| B20 | Human immunodeficiency virus [HIV] disease resulting in infectious and parasitic diseases |
| B21 | Human immunodeficiency virus [HIV] disease resulting in malignant neoplasms |
| B22 | Human immunodeficiency virus [HIV] disease resulting in other specified diseases |
| B24 | Unspecified human immunodeficiency virus [HIV] disease |
| Z21 | Asymptomatic human immunodeficiency virus [HIV] infection status |

One point was added to the total score of the Charlson index for each decade after the age of 50 years:

50 to 59: 1 point, 60 to 69: 2 points, 70 to 79: 3 points, 80 to 89: 4 points, >90: 5 points.

• CHA<sub>2</sub>DS<sub>2</sub>-VACs score: The CHA<sub>2</sub>DS<sub>2</sub>-VASc score will be used to analyze the effect of stratification of the risk of stroke. CHA<sub>2</sub>DS<sub>2</sub>-VASc scores range from 0 to 9. ICD-10 diagnostic codes for each component of the index when applicable:

**C:** I11.0, I13.0, I13.2, I50

Score 1 point

| ICD-10 | Description |
|---|---|
| I110 | Hypertensive heart disease with (congestive) heart failure |
| I130 | Hypertensive heart and renal disease with (congestive) heart failure |
| I132 | Hypertensive heart and renal disease with both (congestive) heart failure and renal failure |
| I50 | Heart failure |

#### **H:** I10, I11, I12, I13, I15

Score 1 point

| ICD-10 | Description |
|--------|--------------------------------------|
| I10 | Essential (primary) hypertension |
| I11 | Hypertensive heart disease |
| I12 | Hypertensive renal disease |
| I13 | Hypertensive heart and renal disease |
| I15 | Secondary hypertension |

### A: Age $\geq$ 75 years

Score 2 points

#### **D:** E10 a E14

Score 1 point

| ICD-10 | Description |
|--------|-----------------------------------------|
| E10 | Insulin-dependent diabetes mellitus |
| E11 | Non-insulin-dependent diabetes mellitus |
| E12 | Malnutrition-related diabetes mellitus |
| E13 | Other specified diabetes mellitus |
| E14 | Unspecified diabetes mellitus |

#### **S2:** G45.0, G45.1, G45.2, G45.3, G45.8, G45.9

Score 2 points

| ICD-10 | Description |
|--------|------------------------------------------------------------------|
| G450 | Vertebro-basilar artery syndrome |
| G451 | Carotid artery syndrome (hemispheric) |
| G452 | Multiple and bilateral precerebral artery syndromes |
| G453 | Amaurosis fugax |
| G458 | Other transient cerebral ischaemic attacks and related syndromes |
**V:** 126, 182, 121- 125, 165, 170- 172, 173.1, 173.8, 173.9, 179.0, 179.2, K55.1, K55.8, K55.9, Z95.8, Z95.9

Score 1 point

| ICD-10 | Description |
|---|---|
| I26 | Pulmonary embolism |
| I82 | Other venous embolism and thrombosis |
| I21 | Acute myocardial infarction |
| I22 | Subsequent myocardial infarction |
| I23 | Certain current complications following acute myocardial infarction |
| I24 | Other acute ischaemic heart diseases |
| I25 | Chronic ischaemic heart disease |
| I65 | Occlusion and stenosis of precerebral arteries, not resulting in cerebral infarction |
| I70 | Atherosclerosis |
| I71 | Aortic aneurysm and dissection |
| I72 | Other aneurysm |
| I731 | Thromboangiitis obliterans [Buerger] |
| I738 | Other specified peripheral vascular diseases |
| I739 | Peripheral vascular disease, unspecified |
| I790 | Aneurysm of aorta in diseases classified elsewhere |
| 1792 | Peripheral angiopathy in diseases classified elsewhere |
| K551 | Chronic vascular disorders of intestine |
| K558 | Other vascular disorders of intestine |

**A:** Age 64-74 years

Score I point

Sc: Sex category (female)

Score 1

• **HASBLED score:** The HAS-BLED score will be used to analyze the risk of bleeding. The modified HAS-BLED score ranges from 0 to 8. ICD-10 diagnostic codes for each component of the index when applicable:

**H:** I10, I11, I12, I13, I15

Score 1 point

| ICD-10 | Description |
|--------|--------------------------------------|
| I10 | Essential (primary) hypertension |
| I11 | Hypertensive heart disease |
| I12 | Hypertensive renal disease |
| I13 | Hypertensive heart and renal disease |
| I15 | Secondary hypertension |

**A:** N03.2, N03.3, N03.4, N03.5, N03.6, N03.7, N05.2, N05.3, N05.4, N05.5, N05.6, N057, N18-N19, N25.0, Z49.0, Z49.2, Z94.0, Z99.2

Score 1 point

| ICD-10 | Description |
|--------|--------------------------------------------------------|
| N032 | Diffuse membranous glomerulonephritis |
| N033 | Diffuse mesangial proliferative glomerulonephritis |
| N034 | Diffuse endocapillary proliferative glomerulonephritis |
| N035 | Diffuse mesangiocapillary glomerulonephritis |
| N036 | Dense deposit disease |
| N037 | Diffuse crescentic glomerulonephritis |
| N052 | Diffuse membranous glomerulonephritis |
| N053 | Diffuse mesangial proliferative glomerulonephritis |
| N054 | Diffuse endocapillary proliferative glomerulonephritis |
| N055 | Diffuse mesangiocapillary glomerulonephritis |
| N056 | Dense deposit disease |
| N057 | Diffuse crescentic glomerulonephritis |
| N18 | Chronic renal failure |
| N19 | Unspecified renal failure |
| N250 | Renal osteodystrophy |
| Z490 | Preparatory care for dialysis |
| Z492 | Other dialysis |
| Z940 | Kidney transplant status |
| Z992 | Dependence on renal dialysis |

# A: B18, I85, I86.4, I98.2, K70, K71.1,K71.3, K71.4, K71.5, K71.7, K72.1, K72.9, K73, K74, K76.0, K76.2, K76.3, K76.4, K76.5, K76.6, K76.7, K76.8, K76.9, Z94.4

Score 1 point

| ICD-10 | Description |
|--------|----------------------------------------------------------|
| B18 | Chronic viral hepatitis |
| I85 | Oesophageal varices |
| I864 | Gastric varices |
| I982 | Oesophageal varices in diseases classified elsewhere |
| K70 | Alcoholic liver disease |
| K711 | Toxic liver disease with hepatic necrosis |
| K713 | Toxic liver disease with chronic persistent hepatitis |
| K714 | Toxic liver disease with chronic lobular hepatitis |
| K715 | Toxic liver disease with chronic active hepatitis |
| K717 | Toxic liver disease with fibrosis and cirrhosis of liver |
| K721 | Chronic hepatic failure |
| K729 | Hepatic failure, unspecified |
| K73 | Chronic hepatitis, not elsewhere classified |
| K74 | Fibrosis and cirrhosis of liver |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K762 | Central haemorrhagic necrosis of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K765 | Hepatic veno-occlusive disease |
| K766 | Portal hypertension |
| Z944 | Liver transplant status |

**S:** I64, I69.3, D62, D68.3, D69.8, D69.9, H31.3, H35.6, H43.1, H45.0, H92.2, I23.0, I31.2 *Score 1 point* 

# Apixaban

# B0661148- NON-INTERVENTIONAL STUDY PROTOCOL

# Final, 10 October 2019

| ICD-10 | Description |
|---|---|
| I64 | Stroke, not specified as haemorrhage or infarction |
| I693 | Sequelae of cerebral infarction |
| D62 | Acute posthaemorrhagic anaemia |
| D683 | Haemorrhagic disorder due to circulating anticoagulants |
| D698 | Other specified haemorrhagic conditions |
| D699 | Haemorrhagic condition, unspecified |
| H313 | Choroidal haemorrhage and rupture |
| H356 | Retinal haemorrhage |
| H431 | Vitreous haemorrhage |
| H450 | Vitreous haemorrhage in diseases classified elsewhere |
| H922 | Otorrhagia |
| I230 | Haemopericardium as current complication following acute myocardial infarction |
| I312 | Haemopericardium, not elsewhere classified |

**B:** I60, I61, I62, I85.0, I98.3, J94.2, K22.6, K25.0, K25.2, K25.4, K25.6, K26.0, K26.2, K26.4, K26.6, K27.0, K27.2, K27.4, K27.6, K28.0, K28.2, K28.4, K28.6, K29.0, K62.5, K66.1, K76.2, K92.0, K92.1, K92.2

# Score 1 point

| ICD-10 | Description |
|--------|---------------------------------------------------------------|
| I60 | Subarachnoid haemorrhage |
| I61 | Intracerebral haemorrhage |
| I62 | Other nontraumatic intracranial haemorrhage |
| I850 | Oesophageal varices with bleeding |
| I983 | Oesophageal varices with bleeding, , not elsewhere classified |
| J942 | Haemothorax |
| K226 | Gastro-oesophageal laceration-haemorrhage syndrome |
| K250 | Acute with haemorrhage |
| K252 | Acute with both haemorrhage and perforation |
| K254 | Chronic or unspecified with haemorrhage |
| K256 | Chronic or unspecified with both haemorrhage and perforation |
| K260 | Acute with haemorrhage |
| K262 | Acute with both haemorrhage and perforation |
| K264 | Chronic or unspecified with haemorrhage |
| K266 | Chronic or unspecified with both haemorrhage and perforation |
| K270 | Acute with haemorrhage |
| K272 | Acute with both haemorrhage and perforation |
| K274 | Chronic or unspecified with haemorrhage |
| K276 | Chronic or unspecified with both haemorrhage and perforation |
| K280 | Acute with haemorrhage |
| K282 | Acute with both haemorrhage and perforation |
| K284 | Chronic or unspecified with haemorrhage |
| K286 | Chronic or unspecified with both haemorrhage and perforation |
| K290 | Acute haemorrhagic gastritis |
| K625 | Haemorrhage of anus and rectum |
| K661 | Haemoperitoneum |
| K762 | Central haemorrhagic necrosis of liver |
| K920 | Haematemesis |
| K921 | Melaena |
| K922 | Gastro-intestinal haemorrhage, unspecified |

L: INR

Score 1 point

**E:** Elderly  $\geq$  65 years

Score 1 point

**D:** E24.4, F10, G31.2, G62.1, G72.1, I42.6, K29.2, K85.2, K86.0, T51, Y90.4, Y90.5, Y90.6, Y90.7, Y90.8, Y91.2, Y91.3, Z50.2, Z71.4, Z72.1

1 or 2 point each

| ICD-10 | Description |
|--------|--------------------------------------------------------|
| E244 | Alcohol-induced pseudo-Cushing's syndrome |
| F10 | Mental and behavioural disorders due to use of alcohol |
| G312 | Degeneration of nervous system due to alcohol |
| G621 | Alcoholic polyneuropathy |
| G721 | Alcoholic myopathy |
| I426 | Alcoholic cardiomyopathy |
| K292 | Alcoholic gastritis |
| K852 | Alcohol-induced acute pancreatitis |
| K860 | Alcohol-induced chronic pancreatitis |
| T51 | Toxic effect of alcohol |
| Y904 | Blood alcohol level of 80-99 mg/100 ml |
| Y905 | Blood alcohol level of 100-119 mg/100 ml |
| Y906 | Blood alcohol level of 120-199 mg/100 ml |
| Y907 | Blood alcohol level of 200-239 mg/100 ml |
| Y908 | Blood alcohol level of 240 mg/100 ml or more |
| Y912 | Severe alcohol intoxication |
| Y913 | Very severe alcohol intoxication |
| Z502 | Alcohol rehabilitation |
| Z714 | Alcohol abuse counselling and surveillance |
| Z721 | Alcohol use |

Codes Anatomical Therapeutic Chemical (ATC): B01AC, M01A

• **SMAe-TT<sub>2</sub>R2 score:** The estimation of SAMe-TT<sub>2</sub>R<sub>2</sub> will be performed by adding the following variables:

**Sex (female)** Score 1 point

Age (<60 years) Score 1 point

Medical history (history of more than two of the following: hypertension, diabetes, coronaty artery disease or myocardial infactions, peripheral artery disease, heart failure, stroke; pulmonary, hepatic, or renal disease)

Score 1 point

Treatment (interacting medications, amiodarone ATC-C01BD01) Score 1 point

**Tobacco use** (within 2 years) Score 2 points

Race (non-Caucasian) Score 2 points

Table 2. Baseline variables or possible confounders

| Variable | Opera | ncional definition ICD-10 |
|---|---|---|
| | E10 | Insulin-dependent diabetes mellitus |
| | E11 | Non-insulin-dependent diabetes mellitus |
| Diabetes | E12 | Malnutrition-related diabetes mellitus |
| Diabetes | E13 | Other specified diabetes mellitus |
| | E14 | Unspecified diabetes mellitus |
| | I10 | Essential (primary) hypertension |
| | I10 | Hypertensive heart disease |
| Hypertension | I11<br>I12 | Hypertensive heart disease Hypertensive renal disease |
| Tryper tension | I12 | Hypertensive heart and renal disease |
| | I15 | Secondary hypertension |
| | I63 | Cerebral infarction |
| Ischaemic stroke | Excepto | |
| ischaemic stroke | 164 | Stroke, not specified as haemorrhage or infarctionz |
| | I60 | Subarachnoid haemorrhage |
| Haamarrhagia straka | I61 | Intracerebral haemorrhage |
| Haemorrhagic stroke | I61<br>I62 | Other nontraumatic intracranial haemorrhage |
| | I60 | |
| | | Subarachnoid haemorrhage |
| | I61<br>I62 | Intracerebral haemorrhage |
| | | Other nontraumatic intracranial haemorrhage |
| | S064 | Epidural haemorrhage |
| | S065 | Traumatic subdural haemorrhage |
| | S066 | Traumatic subarachnoid haemorrhage |
| | I850 | Oesophageal varices with bleeding |
| | K250 | Acute with haemorrhage |
| | K252 | Acute with both haemorrhage and perforation |
| | K254 | Chronic or unspecified with haemorrhage |
| | K256 | Chronic or unspecified with both haemorrhage and perforation |
| | K260 | Acute with haemorrhage |
| | K262 | Acute with both haemorrhage and perforation |
| | K264 | Chronic or unspecified with haemorrhage |
| Bleeding | K266 | Chronic or unspecified with both haemorrhage and perforation |
| _ | K270 | Acute with haemorrhage |
| (gastrointestinal | K272 | Acute with both haemorrhage and perforation |
| intracranial, other) | K274 | Chronic or unspecified with haemorrhage |
| | K276 | Chronic or unspecified with both haemorrhage and perforation |
| | K280 | Acute with haemorrhage |
| | K282 | Acute with both haemorrhage and perforation |
| | K284 | Chronic or unspecified with haemorrhage |
| | K286 | Chronic or unspecified with both haemorrhage and perforation |
| | K290 | Acute haemorrhagic gastritis |
| | K625 | Haemorrhage of anus and rectum |
| | K920 | Haematemesis |
| | K921 | Melaena |
| | K922 | Gastro-intestinal haemorrhage, unspecified |
| | D62 | Acute posthaemorrhagic anaemia |
| | H356 | Retinal haemorrhage |
| | H431 | Vitreous haemorrhage |
| | H450 | Vitreous haemorrhage in diseases classified elsewhere |
| | H922 | Otorrhagia |

# Final, 10 October 2019

| Variable | Onone | ocional definition ICD 10 |
|---|---|---|
| variable | Operacional definition ICD-10 | |
| | I312 | Haemopericardium, not elsewhere classified |
| | J942 | Haemothorax |
| | R04 | Haemorrhage from respiratory passages |
| | K661 | Haemoperitoneum |
| | M250 | Haemarthrosis |
| | N02 | Recurrent and persistent haematuria |
| | N938 | Other specified abnormal uterine and vaginal bleeding |
| | N939 | Abnormal uterine and vaginal bleeding, unspecified |
| | N950 | Postmenopausal bleeding |
| | R31 | Unspecified haematuria |
| | R58 | Haemorrhage, not elsewhere classified |
| | T792 | Traumatic secondary and recurrent haemorrhage |
| Systemic embolism | I74 | Arterial embolism and thrombosis |
| • | E244 | Alcohol-induced pseudo-Cushing's syndrome |
| | E52 | Niacin deficiency [pellagra] |
| | G312 | Degeneration of nervous system due to alcohol |
| | G621 | Alcoholic polyneuropathy |
| | G721 | Alcoholic myopathy |
| | I426 | Alcoholic cardiomyopathy |
| Alcohol consumption | K292 | Alcoholic gastritis |
| | K70 | Alcoholic liver disease |
| | K860 | Alcohol-induced chronic pancreatitis |
| | O354 | Maternal care for (suspected) damage to foetus from alcohol |
| | T51 | Toxic effect of alcohol |
| | Z714 | Alcohol abuse counselling and surveillance |
| | Z721 | Alcohol use |
| D : 1 1 | I702 | Atherosclerosis of arteries of the extremities |
| Peripheral | 1708 | Atherosclerosis of other arteries |
| artery disease | 1709 | Generalised and unspecified atherosclerosis |
| | D50 | Iron deficiency anaemia |
| | D51 | Vitamin B12 deficiency anaemia |
| | D52 | Folate deficiency anaemia |
| | D53 | Other nutritional anaemias |
| Anaemia | D55 | Anaemia due to enzyme disorders |
| | D56 | Thalassaemia |
| | D57 | Sickle-cell disorders |
| | D58 | Other hereditary haemolytic anaemias |
| | D59 | Acquired haemolytic anaemia |
| | I110 | Hypertensive heart disease with (congestive) heart failure |
| <b>Congestive</b> heart | I130 | Hypertensive heart and renal disease with (congestive) heart failure |
| failure | I132 | Hypertensive heart and renal disease with both (congestive) heart failure and |
| lanuic | renal fa | |
| | B15 | Acute hepatitis A |
| | B16 | Acute hepatitis B |
| | B17 | Other acute viral hepatitis |
| | B18 | Chronic viral hepatitis |
| | B19 | Unspecified viral hepatitis |
| Renal disease | C22 | Malignant neoplasm of liver and intrahepatic bile ducts |
| | K70 | Alcoholic liver disease |
| | K71 | Toxic liver disease |
| | K72 | Hepatic failure, not elsewhere classified |
| | K73 | Chronic hepatitis, not elsewhere classified |
| | K74 | Fibrosis and cirrhosis of liver |
| <u> </u> | 12/7 | 1 1010010 und On 110010 Of 11001 |

| Variable | Operacional definition ICD-10 | |
|---|---|---|
| | K75 | Other inflammatory liver diseases |
| | K76 | Other diseases of liver |
| | K77 | Liver disorders in diseases classified elsewhere |
| | Z944 | Liver transplant status |
| Myocardial | I21 | Acute myocardial infarction |
| • | I22 | Subsequent myocardial infarction |
| infarction | I252 | Old myocardial infarction |
| | I70 | Atherosclerosis |
| | I71 | Aortic aneurysm and dissection |
| | I731 | Thromboangiitis obliterans [Buerger] |
| | I738 | Other specified peripheral vascular diseases |
| | I739 | Peripheral vascular disease, unspecified |
| Peripheral vascular | I771 | Stricture of artery |
| <u>-</u> | I790 | Aneurysm of aorta in diseases classified elsewhere |
| disease | I792 | Peripheral angiopathy in diseases classified elsewhere |
| | K551 | Chronic vascular disorders of intestine |
| | K558 | Other vascular disorders of intestine |
| | K559 | Vascular disorder of intestine, unspecified |
| | Z958 | Presence of other cardiac and vascular implants and grafts |
| | Z959 | Presence of cardiac and vascular implant and graft, unspecified |
| | G450 | Vertebro-basilar artery syndrome |
| TIA | G458 | Other transient cerebral ischaemic attacks and related syndromes |
| | G451 | Carotid artery syndrome (hemispheric) |
| | G459 | Transient cerebral ischaemic attack, unspecified |
| <b>Coronary</b> artery | 120 | Angina pectoris |
| disease | I21 | Acute myocardial infarction |

#### 7.4. Data Sources

The information that will be used in the study comes exclusively from secondary sources. Two databases will be used to extract the information:

#### 7.4.1. Claim Database

Claim databasee contains all prescriptions of all patients' medications chronologically. From this database, the index date will be established and the diagnosis of NVAF of the patient will be extracted. Similarly, this base will be used to assess the persistence on therapy and treatment patterns (duration of treatment, changes, persistence), pharmacy claim information, demographic information, diagnosis and insurance data.

#### 7.4.2. Medical Record

Of the patients identified from the claim database, information will be extracted from the second database, the medical record, it will serve to characterize patients based on their baseline demographic and clinical characteristics, that is, on the index date. In turn, it contains the main control variables and the information related to the outcomes of interest, stroke and bleeding events.

# 7.5. Study Size

The total population of patients treated with OAC between January 1, 2013 and June 30, 2018 was analyzed in the claim dabtabase. For the purpose of the study, it contains the information of 7,500 patients, once they were verified that they met the inclusion criteria of the study. This means that patients who start warfarin and NOACs would be included within this period. Patients who initiate NOACs within the established period and who have been exposed to warfarin before 2013 will also be included.

#### 7.6. Data Management

The data sources are databases owned by the investigator, he will execute the data management for this study.

# 7.6.1 Electronic Case Report (ECR)

As used in this protocol, the term ECR should be understood to refer to either a paper form or an electronic data record or both, depending on the data collection method used in this study. ECR is required and should be completed for each included patient. The completed original ECRs are the sole property of Pfizer and should not be made available in any form to third parties, except for authorized representatives of Pfizer or appropriate regulatory authorities, without written permission from Pfizer. The party performing medical record review shall ensure that the ECRs are securely stored at the study site in encrypted electronic form and will be password protected to prevent access by unauthorized third parties.

The party performing medical records review has ultimate responsibility for the abstraction of all clinical, safety, and laboratory data entered on the ECRs and any other data collection forms (source documents).

In order to ensure the accurate, complete, consistent, timely enduring of the data, Pfizer and the third party will design and validate the ECR from review of 30 medical records to guarantee the operationalization adequate of the variables, idenfifying alternative coding data available (abbreviatures, synonyms, symbols, units, etc) and setting of the variables following this protocol. From the results of the validation and the standard operating procedures of Pfizer, data magement plan, data review plan, ECR completion instruction and data entry guidelines will be builted to ensure the consistency and accurate of data. and distribuited to different physicians who participate in the abstraction of the data.

The personal responsible to abstract the data will be physicians who will be trained in the abstraction process, use of manuals and ECR. These grupo will be blinded of the objective of the study in order to avoid the reviewer bias. The party will responsible to conduct and record this activity.

Likewise, the party execute monitoring of tha data which will be follow the guidelines described in the data review plan and data quality control plan as required by the Pfizer policy. Finally, the concordance of the abstracters, the intrarater and interrater reliability, will be measure for cohens kappa and interclass correlation, respectively.

#### 7.6.2 Record Retention

To enable evaluations or inspections/audits from regulatory authorities or Pfizer, third party responsible for performing medical record review agrees to keep all study-related records, including the identity of all participating patients (sufficient information to link records, e.g., ECRs and medical records), ECR file, safety reporting forms, source documents, detailed records of treatment disposition, and adequate documentation of relevant correspondence (e.g., letters, meeting minutes, and telephone call reports). The records should be retained by third party responsible for performing medical record review according to local regulations or as specified in the vendor contract, whichever is longer. Third party responsible for performing medical record review must ensure that the records continue to be stored securely for so long as they are retained.

If third party responsible for performing medical record review becomes unable for any reason to continue to retain study records for the required period, Pfizer should be prospectively notified. The study records must be transferred to a designee acceptable to Pfizer.

Study records must be kept for a minimum of 15 years after completion or discontinuation of the study, unless third party responsible for performing medical record review and Pfizer have expressly agreed to a different period of retention via a separate written agreement. Record must be retained for longer than 15 years if required by applicable local regulations.

The third party responsible for performing medical record review obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

#### 7.6.3 Patient Identification

The Investigators will identify patients from the claim database, initially, in this database the type of therapy with any of the OACs will be verified, and then that they meet the inclusion criteria of the study.

#### 7.6.4 Collection of Information

For the analysis of the data, the statistical package Statistical Package for the Social Sciences (SPSS) Statistics, version 26.0 (IBM, US) for Windows will be used.

Data collection will be performed by healthcare providers following a data collection template developed in Microsoft Excel. For the purpose of unifying criteria and concepts, the template will be parametrized according to the possible responses or options for each variable, which will be defined by the medical expertise, information availability and published clinical studies. The template will be then validated according to a pilot testing of 20 randomly selected clinical charts.

Data collection will be performed after verifying the inclusion and exclusion criteria by the investigation staff. Firstly, the data regarding demographic data and delivery of the medications of interest to the patients meeting the criteria will be reviewed and collected. Subsequently, the electronic medical chart will be reviewed for collecting the clinical data will be identified.

In order to ensure protection of the patient's personal data and maintain high confidentiality and protection of the personal data according to the corporative policy 404 on *Protecting the Privacy of Personal Data*, the vendor will not transfer the collected database.

Pfizer will monitor the vendor to ensure the protection of the patient's personal data.

#### 7.6.5 Database Retention

The Principal Investigator will store the database, adverse event reports and relevant correspondence securely to prevent unauthorized personnel from accessing the information.

# 7.7 Data Analysis

This type of analysis is descriptive and explanatory, as it depends largely on the sample size. Continuous variables will be presented as means, standard deviation or other measures of central tendency or position, while categorical variables will be presented as frequencies and percentages.

Regarding bivariate analyses of continuous variables with normal behavior, the Student's t test will be performed. In case of presenting non-normal behavior, the Mann-Withney test will be used. For variables that are continuous with several categories, analysis of variance (ANOVA) will be assessed. In the event of presenting a non-normal behavior, the multivariate analysis of

variance (MANOVA) test will be carried out. For categorical variables, the X2 test will be used.

Exploratory analyses based on sample size:

The cumulative incidence of clinical outcomes (Stroke/ systemic embolism and major bleeding) will be calculated throughout the study period, from which the incidence or survival curves will be derived using the Kaplan Meier method. Incidence of events will be explored in clinically relevant subgroups based on sample size.

For the execution of the analysis, CCI and change of treatment, and missing treatments are considered as censures. Treatment comparison will be not conducted.

A similar analysis will be performed for the group of patients who have not presented stroke/ systemic embolism or major bleeding events to estimate the time for change of treatment.

In the independent variables, the significance will be analyzed, as a level of statistical significance p < 0.05.

# 7.7.1 Missing Data Management

There will be no imputation or replacement of missing data. All analyses will be conducted on observed cases.

# 7.8 Quality Control

The Principal Investigator or his designee will validate the database constructed, based on the information collected, and they will verify the following:

- Review of illogical data or outliers.
- Verification of conflicting data.
- Review of very high response percentages, such as "unknown" or "not available data"
- Verification of the accuracy of the data collected compared to the source documents
- Report of adverse events (AE)

#### 7.9 Limitations of the research methods

This study, as other observational studies, has some limitations; these are the result of the type of study and the source of information used. It is possible that there is some misclassification of the diagnoses of patients with NVAF as in turn in the diagnoses of the outcomes. For example, in the medical record, it is possible for the Investigator to use indirect information or to relate some type of approximation to obtain the variable or information of interest or to perform. Although this is a risk, the presence has been mitigated through a clear definition of the outcomes and with the case report format, which allows the Investigator to extract the relevant information only.

As for the claim database, a limitation is that prescription does not indicate whether the patient actually took the therapy as prescribed in both dosage and frequency.

On the other hand, this study will not obtain information related to hospitalizations of patients during the follow-up period; therefore, in the event of having any during this period it will not be known if the patient continued therapy. It is worth noting that these types of limitations are not differential among the cohorts of therapies to assess.

In spite of the limitations previously described, this information is very valuable, especially because it allows linking the claim information of medications with the medical records of each patient, providing a large sample size with a significant number of variables.

#### 7.10 Other aspects

Not applicable

#### 8 PROTECTION OF STUDY SUBJECTS

#### 8.1 Patient Information

All parties will comply with all applicable laws, including those relating to the implementation of organizational and technical measures to ensure the protection of patients' personal data. Such measures will include the omission of the patient's name, or other directly identifiable data in reports, publications or other means of dissemination, except when required by the current legislation.

Patient personal data will be stored in the third party research location in an encrypted electronic form and will be password protected to ensure that only authorized study personnel have access. Audifarma will implement the appropriate technical and organizational measures to ensure that personal data may be recovered in the event of a disaster. In the event of a possible violation of personal data, Audifarma will be responsible for determining if there has been a violation of personal data and, if so, providing notifications of violation as required by law.

To protect the rights and freedoms of natural persons with respect to the processing of personal data, when the study data is compiled to be transferred to Pfizer and other authorized parties, any patient's name will be removed and replaced by a unique and specific numerical code. All other identifiable data transferred to Pfizer or other authorized parties will be identified with this unique and specific patient's code. In the event of data transfer, Pfizer will maintain high standards of confidentiality and protection of patients' personal data in accordance with the applicable Audifarma and privacy laws.

#### **8.2 Patient Consent**

As this study does not involve data subject to privacy laws according to applicable legal requirements, obtaining informed consent from patients by Pfizer is not required.

# 8.3 Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

It is the responsibility of the Investigator to have a prospective approval of the study protocol, the protocol amendments, and other relevant documents (for example, recruitment advertisements), if applicable, from the IRB/IEC. All correspondence with the IRB/IEC must be kept in the Investigator's file. Copies of IRB/IEC approvals must be sent to Pfizer.

The study will be evaluated by the Bioethics Committee of the Technological University of Pereira in the category of risk-free research. The principles of confidentiality of the information established by the Declaration of Helsinki will be followed, in accordance with Resolution No. 8430 of 1993 of the Ministry of Health of Colombia. Once you have the support from the committee, the HMO will give authorization to access the medical records.

# 8.4 Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA), Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR).

# 9 MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

The safety reporting language below is applicable to Research staff with oversight of electronic medical records in this study (Human review of unstructured data):

This study protocol requires human review of patient-level unstructured data; unstructured data refer to verbatim medical data, including text-based descriptions and visual depictions of medical information, such as medical records, images of physician notes, neurological scans, X-rays, or narrative fields in a database. The reviewer is obligated to report AE with explicit attribution to any Pfizer drug that appear in the reviewed information (defined per the patient population and study period specified in the protocol). Explicit attribution is not inferred by a temporal relationship between drug administration and an AE, but must be based on a definite statement of causality by a healthcare provider linking drug administration to the AE.

The requirements for reporting safety events on the non-interventional study (NIS) adverse event monitoring (AEM) Report Form to Pfizer Safety are as follows:

- All serious and non-serious AEs with explicit attribution to **any Pfizer drug** that appear in the reviewed information must be recorded on the ECR and reported, within 24 hours of awareness, to Pfizer Safety using the NIS AEM Report Form.
- Scenarios involving drug exposure, including exposure during pregnancy, exposure during breast feeding, medication error, overdose, misuse, extravasation, lack of efficacy and occupational exposure associated with the use of a Pfizer product must be reported, within 24 hours of awareness, to Pfizer Safety using the NIS AEM Report Form.

For these adverse events with an explicit attribution or scenarios involving exposure to a Pfizer product, the safety information identified in the unstructured data reviewed is captured in the Event Narrative section of the report form, and constitutes all clinical information known regarding these AEs. No follow-up on related AEs will be conducted.

All research staff members must complete the following Pfizer training requirements:

"YRR Training for Vendors Working on Pfizer Studies (excluding interventional clinical studies and non-interventional primary data collection studies with sites/investigators)".

These trainings must be completed by research staff members prior to the start of data collection. All trainings include a "Confirmation of Training Certificate" (for signature by the trainee) as a record of completion of the training, which must be kept in a retrievable format. Copies of all signed training certificates must be provided to Pfizer.

# 10 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable Competent Authority in any area of the world, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study patients against any immediate hazard, and of any serious breaches of this NI study protocol that the investigator becomes aware of.

The results will be published in an indexed journal and presented at an international congress according to the availability of the results.

#### 11. REFERENCES

- 1. Molteni M, Polo Friz H, Primitz L, Marano G, Boracchi P, Cimminiello C. The definition of valvular and non-valvular atrial fibrillation: results of a physicians' survey. Europace. 2014;16:1720–5.
- 2. Lip GYH, Nieuwlaat R, Pisters R, Lane DA, Crijns HJGM. Refining Clinical Risk Stratification for Predicting Stroke and Thromboembolism in Atrial Fibrillation Using a Novel Risk Factor-Based Approach. Chest [Internet]. 2010 Feb 1 [cited 2019 Jun 25];137(2):263–72. Available from: https://linkinghub.elsevier.com/retrieve/pii/S0012369210600670
- 3. Olesen J, Lip G, Lindhardsen J, Lane D, Ahlehoff O, Hansen M, et al. Risks of thromboembolism and bleeding with thromboprophylaxis in patients with atrial fibrillation: A net clinical benefit analysis using a 'real world' nationwide cohort study. Thromb Haemost [Internet]. 2011 Nov 29 [cited 2019 Jun 25];106(10):739–49. Available from: http://www.thieme-connect.de/DOI/DOI?10.1160/TH11-05-0364
- 4. Hernández Olmedo M, Suárez Fernández C. Avances en el tratamiento anticoagulante de la fibrilacion auricular. Med Clin (Barc). 2014 Sep;En prensa.
- 5. Banerjee A, Lane DA, Torp-Pedersen C, Lip GYH. Net clinical benefit of new oral anticoagulants (dabigatran, rivaroxaban, apixaban) versus no treatment in a 'real world' atrial fibrillation population: A modelling analysis based on a nationwide cohort study. Thromb Haemost [Internet]. 2012 Nov 22 [cited 2019 Jun 25];107(03):584–9. Available from: http://www.thieme-connect.de/DOI/DOI?10.1160/TH11-11-0784
- 6. Aurachán Torres SA, Ayala Copete AM, Patiño Hermández D, Rios Zuluaga JD, García Peña ÁA, Cano Gutiérrez CA. Riesgo diferencial de hemorragia intracraneana en pacientes con fibrilación auricular no valvular con el uso de nuevos anticoagulantes orales vs. warfarina. Revisión sistemática de la literatura y análisis de subpoblaciones. Univ Médica [Internet]. 2017 Aug 31 [cited 2019 Jun 25];58(2). Available from: http://revistas.javeriana.edu.co/index.php/vnimedica/article/view/19887
- 7. Pinto DA, Sánchez-Vallejo CA, López Pedraza A, Vergara EP, Sáenz ÓA, González F, et al. Descripción de los pacientes con fibrilación auricular no valvular que ingresan al servicio de urgencias. Rev Colomb Cardiol [Internet]. 2016 Jul 1 [cited 2019 Jun 25];23(4):270–6. Available from: https://www.sciencedirect.com/science/article/pii/S0120563315001989
- 8. Nguyen TN, Hilmer SN, Cumming RG. Review of epidemiology and management of atrial fibrillation in developing countries. Int J Cardiol. 2013 Sep;167(6):2412–20.
- 9. Rosselli D, Rodríguez AJ, García ÁA, Rueda JD. Prevalencia de fibrilación auricular en un hospital universitario colombiano. Rev Colomb Cardiol. 2013;20(6):383–5.

# 8. LIST OF TABLES

| Table 1. Table of Variables | 18 |
|-----------------------------------------------------|----|
| Table 2. Baseline variables or possible confounders | 41 |
| 9. LIST OF FIGURES | |
| Figure 1. Study Design | 15 |

Figure 2. Inclusion of Patients ......16

# ANNEX 1. LIST OF STAND ALONE DOCUMENTS

None

# ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable.

# **ANNEX 3. ADDITIONAL INFORMATION**

Not applicable.